CLINICAL TRIAL: NCT00851006
Title: Adjunctive Creatine Treatment for Adolescent Females With Major Depressive Disorder Who Are Non-Responders to Fluoxetine or Escitalopram: A Magnetic Resonance Spectroscopy Study
Brief Title: Creatine Treatment for Female Adolescents With Depression Who Are Non-Responders to Fluoxetine or Escitalopram
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: AlzChem, LLC (Industry)
Responsible Party: Principal Investigator, Douglas Kondo, MD, MD, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 33465
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Females; Adolescents
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-Label Creatine (Experimental): Creatine Monohydrate 4 grams daily by mouth
  Interventions: Drug: Creatine Monohydrate

INTERVENTIONS:
Drug: Creatine Monohydrate — Creapure brand of creatine monohydrate
  Other Names: Creapure

SUMMARY:
The purpose of this study is to see if creatine, which is a naturally occurring chemical in the body, is effective for treating Major Depressive Disorder (MDD) in female teenagers. Creatine may have effects of interest in the brain. The reason for the MRI component of this study is to learn about new ways to see inside the brain. The investigators will use magnetic fields and radio waves to look at the brain and chemicals in the brain. The investigators hope that this technique will have medial use in the future.

The primary hypothesis of the study is that oral creatine supplementation will have a beneficial effect as adjunctive therapy in female adolescents with MDD who are non-responders to an adequate trial of the SSRIs Fluoxetine or Escitalopram.

DETAILED DESCRIPTION:
This is an open-label clinical trial of the investigational drug creatine, for augmentation treatment of female adolescents with Major Depressive Disorder (MDD) who have failed to respond to first-line treatment with Fluoxetine or Escitalopram. Widely used by high school and college athletes in the U.S., creatine is an over-the-counter nutritional supplement with annual sales of more than $200 million. Studies in animals show that creatine improves the performance of female rats in the Porsolt Forced Swim test, which is used to predict the efficacy antidepressant compounds. Human neuroimaging studies indicate that patients with MDD have abnormal levels of high-energy phosphate metabolites in brain, primarily adenosine triphosphate (ATP) and phosphocreatine. Research has also shown that creatine supplementation induces changes in these high-energy phosphate metabolites that are associated with a positive response to antidepressants. For the proposed study, ten female adolescents between the ages of 13-18 with MDD will be recruited for participation in an open-label trial of creatine. Participants with depression will have unremitted MDD despite treatment with Fluoxetine at a dose > 40mg daily for > 4 weeks or Escitalopram at a dose of > 10 mg daily for > 4 weeks. Depressed participants will be treated with oral creatine 4gm daily for eight weeks, and will continue to take Fluoxetine or Escitalopram as prescribed. In addition, ten healthy control participants with no history of psychiatric or substance abuse disorder will be recruited. No treatment will be administered to the control participants. The primary outcome measure will be the Children's Depression Rating Scale (CDRS-R), which was used in the Treatment for Adolescents with Depression Study (TADS) clinical trial (March et al., JAMA 2004; 292(7):807-20) and the Treatment of Resistant Depression in Adolescents (TORDIA) study (Brent et al., JAMA 2008;299(8):901-13). All study participants will undergo brain scans at baseline and again after six weeks, with 31-Phosphorus Magnetic Resonance Spectroscopy (31P-MRS). The brain scans will be used to measure high-energy phosphate metabolites in the Anterior Cingulate Cortex (ACC), an anatomical region of the brain that has been implicated in MDD. 31P-MRS is a non-invasive neuroimaging technique that does not expose participants to radiation. At the magnetic field strength utilized (3T), magnetic resonance imaging is FDA-approved and has no known adverse effects. The research team will use data from 31P-MRS scans to compare levels of high-energy phosphate metabolites in MDD participants vs. healthy controls. In addition, comparison of pre- and post-treatment metabolite levels will be conducted in the MDD participants. The primary hypothesis of the study is that oral creatine will show efficacy as an augmentation treatment for female adolescents with MDD whose depression has not responded to Fluoxetine or Escitalopram. Secondary hypotheses include the following: adolescents with treatment-resistant MDD will show differences at baseline from healthy controls in high-energy phosphate metabolites in the ACC; and that brain scans in depressed adolescents who respond to creatine will show normalization of high-energy phosphate metabolites in the ACC.

ELIGIBILITY:
Inclusion Criteria for Major Depressive Disorder Participants:

* Participants must meet DSM-IV-TR criteria for Major Depressive Disorder, with current mood state depressed for ≥ 2 weeks.
* Participants must be females
* Participants must be between the age of 13 and 18 years.
* Participants must have had an adequate trial of fluoxetine, defined as a trial of ≥ 8 weeks of treatment, with a dose of ≥ 40mg daily for ≥ 4 weeks. If the participant had a trial of 40mg daily and was unable to tolerate it, a dose of 20mg for ≥ 8 weeks is acceptable; OR
* Participants must have had an adequate trial of escitalopram, defined as a trial of ≥ 8 weeks of treatment, with a dose of ≥ 20 mg daily for ≥ 4 weeks. If the participant had a trial of 20 mg daily and was unable to tolerate it, a dose of 10 mg for ≥ 8 weeks is acceptable.
* Participants must have a CDRS-R score of ≥ 40 and a CGI-S score of ≥ 4.
* Participants must be able to give informed consent or assent, and where applicable, parent(s)/guardian(s) must be able to give informed permission for study participation.

Inclusion Criteria for Healthy Control Participants:

* Participants must be females
* Participants must be between the age of 13 and 18 years.
* Participants must not meet DSM-IV-TR diagnostic criteria for a psychiatric or substance abuse disorder.
* Participants must be able to give informed consent or assent and, where applicable, parent(s)/guardian(s) must be able to give informed permission for study participation.

Exclusion Criteria for Treatment-Resistant Major Depressive Disorder Participants:

* Unstable co-morbid medical, neurological or psychiatric disorder.
* Pre-existing renal disease.
* Proteinuria or microalbuminuria.
* Pregnant females, nursing mothers, or females of childbearing potential who are unable or unwilling to practice birth control during the study. Participants who are of child-bearing potential must have a negative urine pregnancy test before each MRI/MRS brain scan.
* High risk for suicidal behavior, homicidal behavior or self-harm.
* Adolescents who are unlikely to be able to comply with the study protocol.
* DSM-IV-TR criteria for current substance abuse or substance dependence, with the exception of nicotine abuse or dependence.
* Contraindication to MRI/MRS brain scans, such as ferromagnetic implants or claustrophobic anxiety.
* Documented or suspected history of intellectual disability (Full-Scale I.Q. < 70).
* History of hypersensitivity to creatine monohydrate.

Exclusion Criteria for Healthy Controls:

* Clinically significant psychiatric or substance abuse disorder.
* Unstable medical or neurological illness.
* Pregnancy, due to the unknown effects of MRI/MRS scanning on a developing fetus.
* Females of childbearing potential who are unable or unwilling to practice contraception during the study.
* Positive urine pregnancy test.
* Contraindication to MRI/MRS scanning, such as ferromagnetic implant or claustrophobic anxiety.
* Documented or suspected history of mental retardation (Full-Scale I.Q. < 70).

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2009-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas G Kondo, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Kondo DG, Hellem TL, Sung YH, Kim N, Jeong EK, Delmastro KK, Shi X, Renshaw PF. Review: magnetic resonance spectroscopy studies of pediatric major depressive disorder. Depress Res Treat. 2011;2011:650450. doi: 10.1155/2011/650450. Epub 2010 Oct 4. PMID 21197097
- [Result] Kondo DG, Sung YH, Hellem TL, Fiedler KK, Shi X, Jeong EK, Renshaw PF. Open-label adjunctive creatine for female adolescents with SSRI-resistant major depressive disorder: a 31-phosphorus magnetic resonance spectroscopy study. J Affect Disord. 2011 Dec;135(1-3):354-61. doi: 10.1016/j.jad.2011.07.010. Epub 2011 Aug 9. PMID 21831448
- See also: University of Utah Brain Institute Website — http://UtahBrain.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Creatine Treatment: Participants with MDD were treated with fixed-dose Creapure® brand of creatine (AlzChem LLC, Trostberg, Germany) 4 g by mouth daily for 8 weeks.
- Healthy Control Group: Only 31P MRS brain scans were used from healthy individuals. HC group were not treated.
Period: Overall Study
Arm/Group | Open Label Creatine Treatment | Healthy Control Group
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Open Label Creatine Treatment: Participants with MDD were treated with fixed-dose Creapure® brand of creatine (AlzChem LLC, Trostberg, Germany) 4 g by mouth daily for 8 weeks. Inclusion criteria were: females 13-18 years of age with a primary diagnosis of MDD. All participants were Caucasian females.
Arm/Group | Open Label Creatine Treatment
Number analyzed (Participants) | 7
Age, Continuous [Mean (Full Range); unit: years]
  Age | 15.6 [14 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Children's Depression Rating Scale (CDRS-R) [Reference: Poznanski EO et al. Preliminary Studies of the Reliability and Validity of the Children's Depression Rating Scale. J Am Acad Child Psychiatry. 1984 Mar;23(2):191-7.]
Description: The CDRS-R is a 17-item scale, with items ranging from 1 to 5 or 1 to 7 (possible total score from 17 to 113), rated by a clinician via interviews with the child or parent. Scores ≥40 are indicative of depression, whereas scores ≤28 is often used to define remission
Time Frame: 8 weeks
Population: This outcome measure was not assessed in the "Healthy Controls". Only subjects in treatment group were evaluated with CDRS-R and received scores.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Open Label Creatine Treatment: The seven subjects who completed the protocol received creatine in the 1-8 week interval. Creatine was initiated at week 0 and terminated at week 8.
Arm/Group | Open Label Creatine Treatment
Number analyzed (Participants) | 7
Units on a scale
  Baseline | 69 (9.69)
  After 8 week Creatine treatment | 30.6 (8.5)

2. Secondary Outcome: 31-phosphorus Magnetic Resonance Spectroscopy Phosphocreatine Metabolite
Description: Phosphocreatine Metabolite is a phosphorylated creatine molecule that plays a role in the production of the energy in the body. Phosphocreatine (PCr) metabolite was quantified by calculating the ratio of PCr over total phosphorus resonance from 31-Phosphorus Magnetic Resonance Spectroscopy.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: ratio of PCr and total phosphorus
Groups:
- Open Label Creatine Treatment: MDD participants' 31P MRS scans were performed prior to the first dose of creatine, and repeated following 8 weeks of treatment.
  Participants were treated with fixed-dose Creapure® brand of creatine (AlzChem LLC, Trostberg, Germany) 4 g by mouth daily for 8 weeks.
- Healthy Control Group: 6 healthy controls returned 8 weeks later for a follow-up scan. HC group did not receive any treatment.
Arm/Group | Open Label Creatine Treatment | Healthy Control Group
Number analyzed (Participants) | 7 | 6
ratio of PCr and total phosphorus
  Baseline | 0.1513 (0.0137) | 0.1556 (0.0086)
  After 8 weeks | 0.1610 (0.0165) | 0.1558 (0.0154)

ADVERSE EVENTS:
Groups:
- Open Label Creatine Treatment: There were no serious adverse events were experienced in this study.
- Healthy Control Group: Healthy Control Group did not go through treatment. HC 31P MRS scans were only used for the study.
Arm/Group | Open Label Creatine Treatment | Healthy Control Group
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 7/7 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Creatine Treatment (N=7) | Healthy Control Group (N=6)
Intermittent tremors (Nervous system disorders) | 1 (1) | 0
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0
Respiratory issues (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0
Gastrointestinal issues (Gastrointestinal disorders) | 5 (6) | 0
Headache, flu-like symptoms, epistaxis, allergies (General disorders) | 3 (9) | 0
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No